CLINICAL TRIAL: NCT07075224
Title: Pharmacodynamics of Investigational Medicinal Product (IMP) 08P2002F0 (Fixed Dose Combination of 0.34 % Tropicamide and 2.5 % Phenylephrine Hydrochloride, Eye Drop Solution), a New Ophthalmic Mydriatic Solution in Healthy Volunteers
Brief Title: Pharmacodynamics of a Fixed Dose Combination of 0.34% Tropicamide and 2.5% Phenylephrine Hydrochloride, Eye Drop, Solution
Acronym: SOLMYD-PD
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Unither Pharmaceuticals, France (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: UP-CLI-2023-01; 2024-517456-35-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-30; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Mydriasis
Keywords: Mydriasis; Mydriatics; Phenylephrine; Tropicamide
MeSH Terms: conditions — Mydriasis

STUDY DESIGN:
Intervention Model Description: Open-label, Observer-masked, active-controlled, randomized cross-over phase I/II study in healthy volunteers.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMP 08P2002F0 (Experimental): 1 eye drop. Rinsing will be performed with NaCl 30 min after instillation
  Interventions: Drug: IMP 08P2002F0
- Mydriasert® insert (Active Comparator): 1 insert will be kept onto the eye for one hour. Then Insert is retrieved and rinsing will be performed with NaCl after retrieval of insert (performed after a contact time of 60 min).
  Interventions: Drug: Mydriasert® insert

INTERVENTIONS:
Drug: IMP 08P2002F0 — Fixed combination of 0.34 % tropicamide and 2.5 % phenylephrine Hydrochloride (HCl) Eye drop Solution.
  Arms: IMP 08P2002F0
Drug: Mydriasert® insert — 0.28 mg tropicamide and 5.4 mg phenylephrine hydrochloride
  Arms: Mydriasert® insert

SUMMARY:
The objective of this study is to explore pharmacodynamic effects and safety of IMP 08P2002F0 for dilation of the pupil, a solution combining two mydriatic agents tropicamide and phenylephrine hydrochloride at the concentrations of 0.34% and 2.5% respectively, versus Mydriasert®

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both genders, aged ≥18 at the time of signing the informed consent.
* Healthy volunteers are declared healthy based on medical history, physical examination, ophthalmological examination, Electrocardiogram (ECG), within the stated normal range; a participant with a clinical abnormality or laboratory parameter(s) outside the reference range may be included if the investigator agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures or interpretation..

  3. Females who participate in the study, that are at reproductive age agree to undergo pregnancy tests and to use a highly effective birth control method during the study.

Exclusion Criteria:

* Hypersensitivity to the active substances or to the excipients or related class of the medicinal product. Serious hypersensitivity reactions include angioedema, anaphylaxis and exfoliative skin conditions including Stevens-Johnson syndrome.

  * Clinically significant illness or surgery within four weeks prior IMP administration.
  * Clinically significant ECG abnormalities or vital sign abnormalities (seated systolic blood pressure < 90 or >140 mmHg, seated diastolic blood pressure < 50 or > 90 mmHg or heart rate less than 50 or over 100 bpm) at screening.

History or presence of any clinically significant cardiovascular, pulmonary, hepatobiliary, renal, haematological, gastrointestinal, endocrinologic, immunologic, dermatologic, neurological, psychiatric, metabolic, musculoskeletal, malignant disease or eye disorders as glaucoma or a family history of glaucoma.

* Clinically significant abnormal laboratory values.
* Unwilling to discontinue use of contact lenses on the day of a treatment visit.
* Current active eye disease (i.e. any disease for which topical or systemic ophthalmic medication is necessary). In case of historical eye disease, topical or systemic ophthalmic medication should have been stopped for at least one month before the study.
* Pupillary abnormalities (irregular, very dark iris, iris synechiae, eye movement disorder (e.g. Nystagmus, etc.), dacryocystitis and all other pathologies of tears drainage system.
* Use of any ophthalmic medication except unpreserved artificial tears on the day of a treatment visit.
* History of inflammatory ocular disease (e.g. iritis, uveitis, herpetic keratitis).
* History of ocular trauma, infection or inflammation within the last 3 months.
* Ocular surgery or laser treatment of any kind in the study eye within 3 months.
* Irregularly-shaped pupil secondary to ocular trauma, intraocular surgery or congenital defect.
* History of neurogenic pupil disorder (e.g. Horner's syndrome, third cranial nerve palsy, Adie's pupil, Argyl Robertson syndrome, etc.).
* History of iris surgery of any kind (e.g. iridotomy, iridectomy, coreoplasty).
* History of previous corneal surgery; iris atrophy, traumatic mydriasis or angle recession, chronic or acute uveitis.
* Corneal, epithelial, stromal or endothelial, residual or evolutionary disease (including corneal ulceration and superficial punctuate keratitis).

Pseudoexfoliation, exfoliative syndrome.

* History of closed-angle glaucoma.
* Subjects with narrow angle prone to glaucoma precipitated by mydriatics
* Subject undergoing treatment identified as potentially interacting with the IMP, including antidepressant drugs, beta-blockers, other indirect sympathomimetics, alpha sympathomimetics (oral and/or nasal routes), dopaminergic ergot alkaloids, ergot alkaloid vasoconstrictors, selective MAOI-A, linezolid, and halogenated volatile anesthetics.

  -. Subject planning to receive an MAOI within 3 weeks following the end of the study.
* Subjects who have received non-selective monoamine oxidase inhibitors (MAOIs) within the last 15 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-09-27 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in pupil diameter at 60 minutes from the time of first dose versus baseline, as measured with photo (central reading) | 60 minutes

SECONDARY OUTCOMES:
Time to obtain sufficient mydriasis | 6 hours post dose
  defined as pupil diameter of 7 mm
Proportion of eyes achieving pupil diameter of 6.0 mm or greater | Throughout the 6 hours, at 30 minutes, at 1 hour and 2 hours.
Proportion of eyes achieving pupil diameter of 7.0 mm | Throughout the 6 hours, at 30 minutes, at 1 hour and 2 hours.
Time from baseline to maximal pupil dilation | 6 hours post dose
Change in pupil diameter at other timepoints | At 10 minutes, 20 minutes, 30 minutes, 45 minutes, 60 minutes, 1 hour and 15 minutes, 1 hour and 30 minutes, 2 hours, 2 hours and 30 minutes, 3 hours, 3 hours and 30 minutes, 4 hours, 4 hours and 30 minutes, 5 hours, 6 hours.
Pupil size | At 10 minutes, 20 minutes, 30 minutes, 45 minutes, 60 minutes, 1 hour and 15 minutes, 1 hour and 30 minutes, 2 hours, 2 hours and 30 minutes, 3 hours, 3 hours and 30 minutes, 4 hours, 4 hours and 30 minutes, 5 hours, 6 hours.
Distribution of pupil diameters | At 10 minutes, 20 minutes, 30 minutes, 45 minutes, 60 minutes, 1 hour and 15 minutes, 1 hour and 30 minutes, 2 hours, 2 hours and 30 minutes, 3 hours, 3 hours and 30 minutes, 4 hours, 4 hours and 30 minutes, 5 hours, 6 hours
Subject ocular discomfort | At 10 minutes, 30 minutes, 60 minutes, 1 hour and 30 minutes, 2 hours, and 6 hours post-administration.
  Healthy volunteers will be asked to respond regarding the following ocular signs after instillation of the respective IMP: irritation/burning/stinging, eye dryness, foreign body sensation, blurred vision by "yes" or "no" and to assess the severity by grading 0 = none, 1 = slight, 2 = moderate, 3 = severe, if sign(s) were noted with "yes" A higher score means a worse result.
Percent of Subjects' Study Eyes with Pupil Diameter Returning to Baseline | Throughout the 6 hours, at 3 hours, 4 hours, 5 hours, 6 hours.
Percentage of subjects' study eyes returning to less than or equal to 0.2 mm from baseline pupil diameter | Throughout the 6 hours, at 3 hours, 4 hours, 5 hours, 6 hours.

OTHER OUTCOMES:
Occurrence of Adverse event | Day 10 post dose
Ocular symptoms other than mydriasis | Day 10 post dose

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Ophthalmiatreion Athinon, Athens
  - Iaso Thessalia General Clinic Private Obstetrics S.A., Larissa

IPD SHARING:
Plan to Share IPD: No